| ANKARA BİLKENT CİTY HOSPİTAL | | | | |
|---|---|---|---|---|
| INFORMED CONSENT FORM – MINIMUM REQUIRED INFORMATION | | | | |
| Document No | Initial Publication Date | Revision Date | Revision No | Page |
| KAD-DD-13 | 01.12.2019 | 20.03.2023 | 01 | 1/2 |

Patient Name – Surname:

Date of Birth:

Archive No / Admission No:

Date:

Study Title: How Safe is Minimal Flow Anesthesia in Terms of Infection Risk?

Minimal flow anesthesia helps maintain the cleanliness of the operating room air, reduces the cost of surgery, lowers the carbon footprint, and contributes to environmental protection. This anesthesia technique, which is both financially and ecologically advantageous, offers important benefits for you by humidifying and warming the gases you inhale, helping to protect your lungs, and preserving body temperature more effectively. It also contributes to more natural and comfortable breathing during surgery and helps maintain the protective mechanisms of your respiratory tract against microorganisms.

The aim of our study is to determine whether the increase in humidity and heat resulting from minimal flow anesthesia causes microorganism colonization in the anesthesia circuit components. Previous studies with low-flow anesthesia have not demonstrated colonization, and our study intends to further investigate minimal flow anesthesia.

This medical study will randomly include 140 voluntary participants. Patients will be assigned by sealed envelope method: 70 patients will receive minimal flow anesthesia and 70 patients will receive normal flow anesthesia. During the research, anesthesia follow-up and treatment in accordance with current standards, along with routine interventional procedures, will be performed. Additionally, prior to anesthesia induction, a throat swab will be taken using a sterile swab stick. The samples collected during the study will be analyzed in the microbiology laboratory of our hospital.

There are no anticipated additional risks or discomforts for volunteers in this study. If there is no clinical benefit expected for you from this study, you will be informed of this. Since routine anesthesia practices will be applied, there are no alternative treatment methods or plans specific to this study other than those mentioned in the standard anesthesia consent form.

Participation in the study is voluntary. You may refuse to participate or withdraw from the study at any time without penalty or loss of rights. In addition, your participation may be terminated by your anesthesiologist or surgeon if deemed necessary.

All records that may identify you will be kept confidential and will not be disclosed to the public. Even if the study results are published, your identity will remain confidential. Authorized monitors, auditors, ethics committees, institutional officials, and relevant health authorities may have direct access to your original medical records, but this information will remain confidential. By signing this written informed consent form, you or your legal representative consent to this access.

| PREPARED BY | COORDINATED BY | APPROVED BY |
|----------------------|---------------------|-----------------|
| Unit Quality Officer | Quality Coordinator | Department Head |

| ANKARA BİLKENT CİTY HOSPİTAL | | | | |
|---|---|---|---|---|
| INFORMED CONSENT FORM – MINIMUM REQUIRED INFORMATION | | | | |
| Document No | Initial Publication Date | Revision Date | Revision No | Page |
| KAD-DD-13 | 01.12.2019 | 20.03.2023 | 01 | 2/2 |

If new information arises during the study that may affect your willingness to continue participating, you or your legal representative will be informed in a timely manner.

For more information about the research, your rights, or in the case of any adverse events, you may contact:

Dr. Aysun ERŞEN YÜNGÜL at +90 532 425 85 39

"I have read all the explanations in the informed consent form. Written and verbal information regarding the research titled and described above was provided to me by the physician named below. I understand that I am voluntarily participating in this study and may withdraw at any time, with or without justification."

"I voluntarily agree to participate in this study without any pressure or coercion."

| Participant's Full Name: |
|-----------------------------------------------------|
| Date – Time: |
| Signature: |
| Maria de El Maria |
| Witness's Full Name: |
| Date – Time: |
| Signature: |
| Legal Representative's Full Name (if applicable): |
| Date – Time: |
| Signature: |
| Dhysician Dunyiding Information - Name and Cymrones |
| Physician Providing Information – Name and Surname: |
| Date – Time: |
| Signature: |

| PREPARED BY | COORDINATED BY | APPROVED BY |
|----------------------|---------------------|-----------------|
| Unit Quality Officer | Quality Coordinator | Department Head |